CLINICAL TRIAL: NCT02122523
Title: In Vivo Study to Determine the Efficacy of Sentinel Node Mapping in Patients With Colon Carcinoma Using Near-infrared Laparoscopy
Brief Title: Sentinel Lymph Node (SLN) in Colorectal Carcinoma (CRC) With a Near-infrared (NIR)-Dye
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Amsterdam UMC, location VUmc (Other)
Responsible Party: Principal Investigator, M.Ankersmit, MD, Amsterdam UMC, location VUmc
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SLN
Record Dates: First submitted 2014-03-19; First posted 2014-04-24 (Estimated); Last update posted 2014-04-24 (Estimated); Status verified 2014-04

CONDITIONS: Sentinel Lymph Node; Colorectal Cancer; Metastasis
Keywords: Image guided surgery
MeSH Terms: conditions — Colorectal Neoplasms; Neoplasm Metastasis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- SLN identification with NIR-dye-subserosa injection (Experimental): Near-Infrared (NIR) dye Indocyanin Green (ICG) to identify nodes with a newly developed NIR laparoscope. The investigators compared two different injection techniques; subserosal and submucosal injection.
  Interventions: Procedure: Near-Infrared (NIR) dye Indocyanin Green (ICG)
- SLN identification with NIR-dye-submucosal injection (Active Comparator): Near-Infrared (NIR) dye Indocyanin Green (ICG) to identify nodes with a newly developed NIR laparoscope. The investigators compared two different injection techniques; subserosal and submucosal injection.
  Interventions: Procedure: Near-Infrared (NIR) dye Indocyanin Green (ICG)

INTERVENTIONS:
Procedure: Near-Infrared (NIR) dye Indocyanin Green (ICG)

SUMMARY:
The sentinel lymph node (SLN) procedure is a standard staging technique in several types of cancer. One of the major problems of SLN mapping in colorectal cancer is the lack of an optimal dye and technique for identification of the nodes. In this study the investigators used the Near-Infrared (NIR) dye Indocyanin Green (ICG) to identify nodes with a newly developed NIR laparoscope. The investigators compared two different injection techniques; subserosal and submucosal injection.

Patients planned for a laparoscopic resection of a colorectal carcinoma without distant metastases were included. Dye was injected in the subserosa or submucosa of the bowel. Ten minutes after injection the investigators searched for fluorescent nodes with the NIR laparoscope. Fluorescent nodes were harvested and analyzed by the pathologist using H&E and additional immunohistochemistry.

ELIGIBILITY:
Inclusion Criteria:

* Oral and written Informed Consent (IC)
* Age 18 years and older
* Patients histological or radiological suspicion of colon cancer
* Surgical resection of the tumor
* Regular Pre-operative work-up

Exclusion Criteria:

* Gross lymph node involvement
* Distant metastases
* Advanced disease with invasion of adjacent structures
* Prior colorectal surgery
* Metastatic or T4 disease discovered during intraoperative staging
* Contraindications to laparoscopy
* Rectal cancer
* Allergy to iodine
* Patients at higher risk for anaphylactic reactions

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2013-01; Primary Completion 2014-01 (Actual)

PRIMARY OUTCOMES:
Number of fluorescent lymph nodes | 4 hours

SECONDARY OUTCOMES:
Number of Lymph nodes with metastasis | 4 hours

CONTACTS AND LOCATIONS:
Locations (1):
- VU University Medical Center, Amsterdam, North Holland, Netherlands